CLINICAL TRIAL: NCT07280312
Title: Ultrasound Imaging of Ovarian and Adnexal Lesions
Brief Title: Ultrasound Microvessel Imaging for the Evaluation of Ovarian and Adnexal Lesions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 25-008495; NCI-2025-08526 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 25-008495 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2025-12-02; First posted 2025-12-12 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Female Reproductive System Adnexal Neoplasm; Ovarian Carcinoma; Female Reproductive System Neoplasm; Ovarian Neoplasms; Adnexal Lesion; Ovarian Lesion
MeSH Terms: conditions — Ovarian Neoplasms; Genital Neoplasms, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic (UMI, transvaginal ultrasound) (Experimental): Patients undergo UMI during standard transvaginal ultrasound imaging procedure on study.
  Interventions: Procedure: Transvaginal Ultrasound; Procedure: Ultrasound Microvessel Imaging

INTERVENTIONS:
Procedure: Transvaginal Ultrasound — Undergo transvaginal ultrasound
  Other Names: transvaginal sonography; TVS; TVU
Procedure: Ultrasound Microvessel Imaging — Undergo UMI
  Other Names: 3D Ultrasound Microvessel Imaging; UMI

SUMMARY:
This clinical trial studies how well ultrasound microvessel imaging (UMI) works in evaluating ovarian and adnexal lesions in patients who are scheduled to have surgical treatment for their ovarian or adnexal lesions as part of their clinical care. Ovarian cancer is the most lethal gynecologic malignancy, often diagnosed at an advanced stage. Current diagnostic tools include a blood test (serum cancer antigen 125 [CA125]) and transvaginal ultrasound. However, CA125 has limited diagnostic accuracy and is Food and Drug Administration-approved only for monitoring the return of cancer (recurrence), not for preoperative diagnosis. A key measurement in calculating ovarian and adnexal cancer risk is by looking at increased blood flow, which may suggest a higher risk of cancer developing. However, current ultrasound techniques have limited ability to assess blood flow. A new ultrasound technique, UMI, may have higher sensitivity for detecting small blood vessels compared to traditional ultrasound imaging.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged ≥ 18 years
* Scheduled for surgery for ovarian or adnexal lesions

Exclusion Criteria:

* Prior surgical removal of ovarian or adnexal lesions
* Undergoing neoadjuvant chemotherapy or targeted systemic therapy
* Vulnerable populations, including prisoners, adults lacking capacity to consent, and pregnant women (our study coordinator will ask participants if they are pregnant; if uncertain, a urine pregnancy test will be offered at no cost).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-22 (Actual); Primary Completion 2027-12-17 (Estimated); Study Completion 2029-12-17 (Estimated)

PRIMARY OUTCOMES:
Change in O-RADS score | Baseline
  Ovarian-Adnexal Reporting and Data System (O-RADS) scores will be initially based on B-mode and Doppler imaging (standard of care) obtained prior to surgical treatment. Radiologists will then review ultrasound microvessel imaging (UMI) images and may choose to revise the score. Accuracy of score adjustments will be assessed using final pathology results from the participant's medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Shigao D. Chen, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials